CLINICAL TRIAL: NCT03635502
Title: What Are the Determinants of Explicit and Implicit Motor Imagery Ability in Stroke Patients?: A Controlled Study
Brief Title: What Are the Determinants of Explicit and Implicit Motor Imagery Ability in Stroke Patients?
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Istanbul University (Other); Bakırkoy Dr. Sadi Konuk Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Esma Nur KOLBAŞI, Research Assisstant, Istanbul Medeniyet University
Other Study IDs: IstanbulMU1
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Stroke; Healthy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Group
- Healthy Group

SUMMARY:
Motor imagery (MI) might be described as a dynamic process in which an individual mentally stimulates an action without any overt movement. After stroke, motor imagery ability is impaired and also due to structure of MI, not every stroke patients is able to perform MI. Therefore, the aim of the study is a) to compare both explicit and implicit motor imagery ability (MIA) between patients with stroke and healthy subjects, b) to examine predictive effects of clinical characteristics for MIA after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-80,
* Having a unilateral stroke for the first time and 0-6 months since stroke onset
* 24 points and above in Mini Mental State Examination (MMDM)
* Not having a disease that may interfere with the study such as cardiac diseases, orthopedic conditions,etc.

Exclusion Criteria:

* Multiple strokes
* Sever cognitive dysfunction (<24 points in MMDM)
* Unilateral neglect
* Upper extremity pain that interferes with the study or aggravated with movement
* Visual problems, aphasia or another sequel that might limit the assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients and age, sex, education matched healthy volunteers who meet the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Movement Imagery Questionnaire-3 (MIQ-3) | 15 min
  MIQ-3 evaluates an individual's motor imagery ability in 3 subscales: 1. internal imagery, 2. external imagery, 3. kinesthetic imagery. Each of these scales ranges from 1 to 7 where 1 indicates very hard to see/feel (image) and 7 indicates very easy to see/feel. 12 items are included in the MIQ-3 and every item is scored according to the scales. The higher the score in subscales, the better the results are.
Chaotic Motor Imagery Assessment- Hand Rotation | 20 min
  Hand Rotation is the first component of Chaotic Motor Imagery Assessment. In this measure, 96 drawings of each hand (left and right) from 4 different plane and at 12 different angle are presented to the individuals and then, it is asked to decide whether it is left or right hand. Total test time, total accuracy, total wrong answers, right accuracy, left accuracy, impaired hand and non-impaired hand accuracy is recorded as outcome scores.
Box and Block Test | 5 min
  Box and Block Test is used to calculate mental chronometry (MC) ratio. During the test, patients are asked to carry 15 blocks first physically and then mentally from one box to another. As outcome scores, the time required to carry 15 blocks physically (MET) and mentally (MIT) are recorded. Then MC ratio is calculated with the formula: (MET-MIT)/ MET.
Fugl-Meyer Assessment- Upper Extremity | 10 min
  Upper extremity part of Fugl Meyer Assessment (FMAUE) is used to evaluate patients' motor impairment level. Total motor and sensory scores are recorded. Then, patients are divided into 4 different categories according to their motor impairment level:
  1. 23-31 points: poor upper extremity function,
  2. 32-47 points: limited function,
  3. 48-52 points: notable function, 4.53-66 points: full function.

SECONDARY OUTCOMES:
Motor Activity Log-28 | 5 min
  Turkish version of MAL-28 was used to assess how much (amount of use scale) and how well (how well scale) the patients used their upper extremity in daily life after stroke. These 2 different scales are calculated separately with range of 0-5 points.The higher the points are, the better the patients' situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided